CLINICAL TRIAL: NCT07360847
Title: Profiling Patients With Rotator Cuff Related Shoulder Pain: What Factors Influence Outcomes With Non-operative Care in a Secondary Care Specialist Shoulder Clinic?
Status: Not yet recruiting | Type: Observational
Sponsor: University of Limerick (Other)
Responsible Party: Sponsor
Other Study IDs: 0254 Prospective Cohort Study; GOIPG/2024/2553 (Other Grant/Funding Number: Irish Research Council)
Record Dates: First submitted 2026-01-13; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-12

CONDITIONS: Rotator Cuff Related Shoulder Pain; RCRSP
Keywords: RCRSP; Rotator Cuff Related Shoulder Pain; Non-operative; Prognosis; Prognostic Factor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non-operatively managed Rotator Cuff Related Shoulder Pain patients: Non-operatively managed

SUMMARY:
Shoulder pain from rotator cuff disorders is common, affecting function and quality of life. Many patients in orthopaedic clinics are diagnosed with these conditions. Most do not need surgery and are treated with pain relief and physiotherapy. However, long physiotherapy waitlists cause delays, and some patients do not achieve good outcomes. There is limited evidence to predict who will recover well with non-surgical care.

We propose a cohort study at Croom Orthopaedic Hospital to explore this. Patients assessed as suitable for non-surgical care by the shoulder physiotherapist will provide consent and complete questionnaires on pain, disability, quality of life, and personal factors like age and gender. They will continue with prescribed care and repeat the questionnaires after six months.

This study will identify factors predicting successful outcomes, improving treatment programs to better meet patients' needs. It is funded by the Irish Research Council and led by Professors Karen McCreesh and Rose Galvin, UL, and Mr. Tristan Cassidy, Orthopaedic Consultant. Collaborators include Catriona Foley, shoulder specialist physiotherapist at Croom.

DETAILED DESCRIPTION:
Aims and Objectives The overall aim of the study is to examine the factors associated with the outcome of non-surgical care among a cohort of people referred to a specialist shoulder clinic.

The objectives of the study are as follows:

1. To conduct a prospective cohort study of adults with RCRSP presenting to a secondary care clinic in the mid-west suitable for non-operative management.
2. To determine the association between key patient characteristics (demographics, level of disability, comorbidities, etc) and outcome following physiotherapy management of RCRSP.

Introduction Shoulder pain is the third most common musculoskeletal symptom reported in primary care and has a prevalence of up to 26% in the general population (Rangan et al., 2016). It is a disabling condition, and when symptoms persist, it can impair quality of life, increase psychological distress and reduce the ability to maintain employment (Ackerman et al., 2018). Disorders of the rotator cuff muscle and tendons are the most commonly diagnosed cause of shoulder pain. A strong body of research evidence currently exists recommending non-surgical management (e.g. exercise) as the preferred first-line treatment for rotator cuff disorders (Littlewood et al., 2018). Shoulder surgery is more than twice as expensive as conservative approaches, and more importantly, has not been shown to produce superior outcomes in terms of pain and function compared to no treatment or non-surgical management (Beard et al., 2018, Ryösä et al., 2017, Ketola et al, 2013). Despite this, surgery rates continue to rise (Rangan et al., 2018).

Non-operative management includes the use of analgesia, physiotherapist led exercise and advice, and judicious use of corticosteroid injections (LaFrance et al., 2022). However, many patients are not receiving guideline based care in the primary care setting and are being unnecessarily referred to secondary care (Maxwell et al., 2022). In addition, due to resource constraints, long waiting times exist within primary care physiotherapy negatively impact patient outcomes and increase overall costs of care (Deslauriers et al., 2019). Recent evidence has found that a single advice and education session with a trained physiotherapist followed by a home self-management programme, produced equivalent outcomes to a control intervention of up to six face-to-face physiotherapy session for people with rotator cuff disorders (Marian et al., 2020). A recent systematic review by the research team of this model of care has confirmed this finding applies across a range of musculoskeletal disorders. While this research suggests that a 'less is more' approach can be successful in managing musculoskeletal pain, it is likely that some patient cohorts will require more intensive input, as illustrated in studies of low back where those with higher levels of mental health disorders needed more intensive multi-disciplinary input (Haglund et al., 2019). Therefore, it is important to identify predictors of negative outcomes with non-operative care so that an intervention can be developed which aims to address any modifiable prognostic factors.

A more effective method of education and exercise rehabilitation is required in order to optimise patient outcomes, particularly with our primary care facilities at capacity and patients experiencing long wait times for Physiotherapy referral. Carefully designed and implemented education and exercise rehabilitation programmes have the potential to bridge this gap. Research that is collaborative is vital to ensure education and exercise programmes match the needs of patients with RC disorders in the Mid-west.

Intervention Patients recruited for this study will undergo usual physiotherpy care. This typically involves referral to community physiotherapy.

Conservative management strategies will be provided by CORU registered Physiotherapists. Those non-operative strategies included in "usual care" can include one or more of the following; exercise, education, acupuncture, manual therapy, local injection of steroids or anaesthesia, advice, multidisciplinary input.

Control This prospective cohort study aims to identify prognostic factors associated with functional recovery among adults with rotator cuff related shoulder pain. The effectiveness of specific interventions will not be investigated.

Those prognostic factors being investigated and OCM's must be collected at baseline on initial presentation and again after a period of time deemed suitable to produce clinically significant changes in collected OCM's - 6 months.

We will use the International Classification of Function, Disability and Health to characterise prognostic factors under the domains of Body Structures and Function, Activity Limitations, Participation Restrictions, as well as Personal and Environmental factors.

Methodology The Clinical Specialist physiotherapist will triage patients presenting with RCRSP and identify those for whom non-surgical care is prescribed. The research nurse and PhD student will inform patients about the study and invite them to take part. Participants who consent to the study will complete baseline questionnaires. They will be contacted 6 months later to complete a further set of questionnaires.

In the first month, the team will pilot the data collection software (Qualtrics) and study procedures. In a small cohort of 10 patients, we will examine the feasibility of consenting them to the study in advance of the collection of their baseline characteristic and PROM, and then the actual collection of their baseline characteristic and PROM's. This trial will inform the implementation of the project on a larger scale.

Study Design This prospective cohort study is designed to be pragmatic in nature. The methods described below have been developed based on a review of the international literature (evidence-base), the results of a Systematic Review of the Literature and from the output of meetings with the research team working in the secondary care clinic. This qualitative research will be completed prior to commencing the prospective cohort study. The EQUATOR reporting guidelines will be followed to ensure the standardised conduct and reporting of research.

Analysis Prof Rose Galvin, School of Allied Health will provide expert statistical advice and input. Appropriate descriptive statistics will be used to describe the baseline characteristics of study participants. These will include proportions, percentages, ranges, means and standard deviations and medians and interquartile ranges (where data are not normally distributed).

Multiple logistic regression will be used to examine the influence of a variety of factors in patient outcomes.

Conclusion By collecting data on the patient characteristics and Patient reported outcome measures we can better understand the types of people presenting to secondary care clinic with RCRSP.

By tracking their outcomes over six months, we can better understand what patient characteristics and prognostic factors influence outcomes.

In the future, efforts can be made to target modifiable prognostic factors and modify pathways of care to optimise prognosis.

ELIGIBILITY:
Inclusion Criteria:

Adults Clinically diagnosed Rotator Cuff Related Shoulder Pain (disorder of the rotator cuff muscles and/or sub acromial space).

Being referred to primary care physiotherapy or other non-surgical management.

Exclusion Criteria:

Under 18 Non-rotator cuff related pathologies of the shoulder such as fractures, frozen shoulder, concomitant neck pain.

Person undergoing shoulder surgery. Neither the patient nor carer can communicate in English sufficiently to complete consent or baseline assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults who present to the Specialist Shoulder clinic at Croom Orthopaedic Hospital between January 2026 and January 2027 (inclusive) will be considered eligible for inclusion to the study provided that they meet the inclusion criteria outlined above.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Pain VAS | From enrollment to six month follow up
  Pain level on a scale from 0-10
SPADI | From enrollment to six month follow up
  Shoulder Pain and Disability Index measures a patient's self-perceived pain and functional limitations due to shoulder problems.
WORC | From enrollment to six month follow up
  Western Ontario Rotator Cuff Index measures the impact of rotator cuff conditions on a person's quality of life